CLINICAL TRIAL: NCT05853250
Title: Clinical (Sleep, Pain and Atrial Fibrillation) and Hospital Stay Effects of Reiki and Manual Therapy After Open Heart Surgery
Brief Title: Clinical and Hospital Stay Effects of Reiki and Manual Therapy After Open Heart Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Nancy M. Albert, Ph.D., Associate Chief Nursing Officer, Office of Nursing Research, Principal Investigator of record (Sandy Zampino left Cleveland Clinic), The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 17-184
Record Dates: First submitted 2023-04-11; First posted 2023-05-10 (Actual); Results first posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Coronary Artery Diseases; Valvular Heart Diseases
Keywords: Cardiac surgery; Coronary artery bypass grafting (CABG); Valve surgery; Reiki; Manual therapy
MeSH Terms: conditions — Coronary Artery Disease; Heart Valve Diseases | interventions — Therapeutic Touch; Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: Patients were recruited and enrolled into the study preoperatively. After completing baseline information, they were randomized to the intervention or control group. After surgery they received the group assignment.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Personnel who recruited and enrolled patients preoperatively were not involved in any other component of the study. Surgeons and medical providers did not receive any information about group assignment. Reiki/manual therapy personnel did not collect outcome "survey" data; those that did were not informed of group assignment. Data coming from a database was retrieved by a data analyst who did not receive group assignment information.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reiki/manual therapy (Experimental): Reiki, a Japanese energy-based healing technique, is universal vital energy that flows throughout and encompasses all living forms (Rand, 1991). It is delivered by gentle hand placement either on/slightly above the body by certified Reiki practitioners. In this study, Reiki will be delivered first, for 15 min. and will involve light placement of hands on patients' head, chest, shoulders, hands, knees, and feet (~ 3 minutes to each body part). Manual therapy (MT) includes light effleurage to head and feet (for 5 minutes; ~ 2.5 minutes to each body part) by the Reiki practitioner. MT techniques are defined as light circular stroking movements made with the hands. Reiki and MT will be delivered for 3 consecutive days beginning on the day after endotracheal tube removal. Reiki and MT will be delivered by 4 Reiki practitioners with training at a Level 2+. Reiki and manual therapy was delivered as one intervention. They are not two separate interventions.
  Interventions: Other: Reiki/manual therapy
- Usual care quiet time (No Intervention): All usual care provided pre and post-operative management will continue, uninterrupted; including the 20 minute rest period. The only non-usual care component will be placement of a sign on the door to discourage visitors and providers from entering the room and disturbing the rest period.

INTERVENTIONS:
Other: Reiki/manual therapy — Reiki is delivered by gentle hand placement either on or slightly above the body by certified Reiki practitioners. In this study, Reiki will be delivered first, for 15 minutes and will involve light placement of hands on patients' head, chest, shoulders, hands, knees, and feet (~ 3 minutes to each body part). Manual therapy techniques include light effleurage to head and feet (for 5 minutes; ~ 2.5 minutes to each body part) by the Reiki practitioner who delivered the Reiki therapy.
  Arms: Reiki/manual therapy

SUMMARY:
Reiki is an energy-based healing therapy using light touch. Manual therapy is a technique using light effleurage. These complimentary healing services are utilized to promote relaxation, sleep, improve emotions, and decrease pain; however, more research is required since sample sizes in the literature were small, subjects were generally healthy (not hospitalized), and subjects had multiple medical backgrounds. Only 1 study focused on cardiac surgery patients. We aim to learn if Reiki and manual therapy enhances postoperative clinical outcomes for patients after first time coronary artery bypass graft (CABG) and/or cardiac valve surgery. A randomized, controlled non-blinded study will enroll a sample of a minimum of 272 patient (136 per group), based on a power analysis using the primary outcome. The intervention group will receive usual care plus Reiki and manual therapy, with Reiki delivered first. Total therapies time is 20 minutes. Reiki and manual therapy will be delivered for 3 consecutive days beginning on the day after endotracheal tube removal. The usual care group will receive 20 minutes of uninterrupted rest, which is part of usual postoperative care. Outcomes are depression, anxiety, pain, night time sleep, new onset atrial fibrillation, hospital length of stay, all-cause 30-day hospital readmissions, narcotic drug burden and post-operative complications.

DETAILED DESCRIPTION:
Background: Reiki is an energy-based healing therapy using light touch. Manual therapy is a technique using light effleurage. These complimentary healing services are utilized to promote relaxation, sleep, improve emotions, and decrease pain. After reviewing the Reiki research literature, more research is required since sample sizes were small, subjects were generally healthy (not hospitalized), and subjects had multiple medical backgrounds. Only 1 study focused on cardiac surgery patients. In the current research study, we aim to learn if Reiki and manual therapy enhances postoperative clinical outcomes for patients after first time coronary artery bypass graft (CABG) and/or cardiac valve surgery.

Design and Methods: A randomized, controlled non-blinded study will be used. The sample size (272 total; 136 per group) was based on a power analysis using the primary outcome. The intervention group will receive usual care plus Reiki and manual therapy, with Reiki being delivered first. Hand placements include: head, chest, shoulders, hands, knees, and feet for 15 minutes. Manual therapy will consist of light effleurage to the head and feet for 5 minutes. Total therapies time is 20 minutes. Reiki and manual therapy will be delivered for 3 consecutive days beginning on the day after endotracheal tube removal. The usual care group will receive 20 minutes of uninterrupted rest, which is part of usual postoperative care. There will not be a sham-treatment group, based on previous research findings.

Outcome Measures: depression and anxiety (Brief Symptom Inventory, 12-item self-administered tool); pain (self-reported and recorded in electronic health record by staff nurses as part of usual care -- 0 [no pain] - 10 [worst pain] scale), highest (worst) and lowest (least) pain in the past 24 hours will be assessed; night time sleep (Richards-Campbell Sleep Questionnaire; 5 item self-administered tool)-to be measured at baseline and after the last Reiki/manual therapy treatment or 3 days of usual care; hospital length of stay, all-cause 30-day hospital readmissions (data top be retrieved from a billing database), narcotic drug burden (mean dose) use on postoperative days 3 and 4 (retrieved from electronic medical records), patient characteristics, medical history, surgical procedure, new onset atrial fibrillation and other post-operative complications (retrieved from the Institutional Review Board--approved Cardiothoracic Surgery database).

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Speaks English language and capable of reading and hearing
* Up to 4 "To Come In" patients enrolled per day (2 standard care and 2 intervention group)
* Arrive for surgery from outpatient (home) environment
* Scheduled for surgery (arrives in "To Come In" area) on Monday and Tuesday.
* Lives in one of 6 counties of North East Ohio to ensure access post-discharge hospitalization

Exclusion Criteria:

* History of dementia, cognitive decline, Down's syndrome or other neurologic, psychological or congenital deficiency that impacts ability to make decisions about enrollment
* Severe sight and hearing impairment despite assistive devices
* Cardiac surgery on a Wednesday, Thursday or Friday
* Treated in the hospital prior to the day of surgery
* Prolonged intubation (over 48 hours), or reinsertion of an endotracheal tube during or before the intervention is initiated (will result in intervention withdrawal)
* Sedated due to new onset delirium.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2017-06-26 (Actual); Primary Completion 2019-09-18 (Actual); Study Completion 2020-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Zampino, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Albert NM, Gillinov AM, Lytle BW, Feng J, Cwynar R, Blackstone EH. A randomized trial of massage therapy after heart surgery. Heart Lung. 2009 Nov-Dec;38(6):480-90. doi: 10.1016/j.hrtlng.2009.03.001. Epub 2009 Jun 28. PMID 19944872
- [Background] Anderson PG, Cutshall SM. Massage therapy: a comfort intervention for cardiac surgery patients. Clin Nurse Spec. 2007 May-Jun;21(3):161-5; quiz 166-7. doi: 10.1097/01.NUR.0000270014.97457.d5. PMID 17495551
- [Background] Boitor M, Martorella G, Arbour C, Michaud C, Gelinas C. Evaluation of the preliminary effectiveness of hand massage therapy on postoperative pain of adults in the intensive care unit after cardiac surgery: a pilot randomized controlled trial. Pain Manag Nurs. 2015 Jun;16(3):354-66. doi: 10.1016/j.pmn.2014.08.014. PMID 26025795
- [Background] Borm GF, Fransen J, Lemmens WA. A simple sample size formula for analysis of covariance in randomized clinical trials. J Clin Epidemiol. 2007 Dec;60(12):1234-8. doi: 10.1016/j.jclinepi.2007.02.006. Epub 2007 Jun 6. PMID 17998077
- [Background] Braun LA, Stanguts C, Casanelia L, Spitzer O, Paul E, Vardaxis NJ, Rosenfeldt F. Massage therapy for cardiac surgery patients--a randomized trial. J Thorac Cardiovasc Surg. 2012 Dec;144(6):1453-9, 1459.e1. doi: 10.1016/j.jtcvs.2012.04.027. Epub 2012 Sep 7. PMID 22964355
- [Background] Cutshall SM, Wentworth LJ, Engen D, Sundt TM, Kelly RF, Bauer BA. Effect of massage therapy on pain, anxiety, and tension in cardiac surgical patients: a pilot study. Complement Ther Clin Pract. 2010 May;16(2):92-5. doi: 10.1016/j.ctcp.2009.10.006. Epub 2009 Nov 14. PMID 20347840
- [Background] Doering LV, Moser DK, Riegel B, McKinley S, Davidson P, Baker H, Meischke H, Dracup K. Persistent comorbid symptoms of depression and anxiety predict mortality in heart disease. Int J Cardiol. 2010 Nov 19;145(2):188-192. doi: 10.1016/j.ijcard.2009.05.025. Epub 2009 Jun 2. PMID 19493579
- [Background] Gordon DB, Polomano RC, Pellino TA, Turk DC, McCracken LM, Sherwood G, Paice JA, Wallace MS, Strassels SA, Farrar JT. Revised American Pain Society Patient Outcome Questionnaire (APS-POQ-R) for quality improvement of pain management in hospitalized adults: preliminary psychometric evaluation. J Pain. 2010 Nov;11(11):1172-86. doi: 10.1016/j.jpain.2010.02.012. Epub 2010 Apr 18. PMID 20400379
- [Background] Lee MS, Pittler MH, Ernst E. Effects of reiki in clinical practice: a systematic review of randomised clinical trials. Int J Clin Pract. 2008 Jun;62(6):947-54. doi: 10.1111/j.1742-1241.2008.01729.x. Epub 2008 Apr 10. PMID 18410352
- [Background] MacIntyre B, Hamilton J, Fricke T, Ma W, Mehle S, Michel M. The efficacy of healing touch in coronary artery bypass surgery recovery: a randomized clinical trial. Altern Ther Health Med. 2008 Jul-Aug;14(4):24-32. PMID 18616066
- [Background] Mackay N, Hansen S, McFarlane O. Autonomic nervous system changes during Reiki treatment: a preliminary study. J Altern Complement Med. 2004 Dec;10(6):1077-81. doi: 10.1089/acm.2004.10.1077. PMID 15674004
- [Background] Rand W. (1991). The Healing Touch. First and Second Degree Manual. Vision Publication: Southfield, MI.
- [Background] Richards KC, O'Sullivan PS, Phillips RL. Measurement of sleep in critically ill patients. J Nurs Meas. 2000 Fall-Winter;8(2):131-44. PMID 11227580
- [Background] Society of Thoracic Surgeons. The Society of Thoracic Surgeons Adult Cardiac Surgery Database data collection form version 2.81, April 23,2015. Society of Thoracic Surgeons, www.sts.org. Accessed 09-12-2016.
- [Background] vanderVaart S, Gijsen VM, de Wildt SN, Koren G. A systematic review of the therapeutic effects of Reiki. J Altern Complement Med. 2009 Nov;15(11):1157-69. doi: 10.1089/acm.2009.0036. PMID 19922247
- [Background] Vitale A. An integrative review of Reiki touch therapy research. Holist Nurs Pract. 2007 Jul-Aug;21(4):167-79; quiz 180-1. doi: 10.1097/01.HNP.0000280927.83506.f6. PMID 17627194

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From the "to come in" (TCI) list for first time cardiac surgery patients, data collectors retrieved names and interviewed patients that met criteria for the research study. Patients were also enrolled from the Pre-Cath area. Written informed consent was acquired by patients before initiation of the research study. Study recruitment was from 6/26/17 to 9/10/2019.
Pre-assignment Details: The patient's surgery was canceled or delayed therefore these people either did not sign the informed consent or they signed the informed consent, but because surgery did not happen on the day scheduled, they did not participate in the study.
Period: Overall Study
Arm/Group | Reiki/Manual Therapy | Usual Care Quiet Time
Started | 136 | 136
Completed | 136 | 136
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Reiki/Manual Therapy | Usual Care Quiet Time | Total
Number analyzed (Participants) | 136 | 136 | 272
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.4 (11.9) | 62.0 (12.6) | 62.2 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 33 | 67
  Male | 102 | 103 | 205
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 126 | 124 | 250
  Other race/ethnicity | 10 | 12 | 22
Region of Enrollment [Number; unit: participants]
  United States | 136 | 136 | 272
Payor [Count of Participants; unit: Participants]
  Government (Medicare/Medicaid) + Self Pay | 35 | 40 | 75
  Private + Other Inc | 101 | 96 | 197
Primary Diagnosis [Count of Participants; unit: Participants]
  Cardiac | 95 | 108 | 203
  Congenital | 41 | 28 | 69
BMI [Mean (Standard Deviation); unit: kg/m2] | 28.7 (5.3) | 27.8 (5.2) | 28.2 (5.2)

OUTCOME MEASURES:

1. Primary Outcome: Depression
Description: The Brief Symptom Inventory has a depression dimension that includes 6 items. Participants are asked to consider the "past week" when responding and each item is scored on a 5-point scale, from 0 (not at all) to 4 (extremely). The higher the score, the worse the depression; score range is 0-24.
Time Frame: Pre-operative (baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reiki/Manual Therapy | Usual Care Quiet Time
Number analyzed (Participants) | 136 | 136
score on a scale | 0.31 (0.46) | 0.42 (0.58)

2. Primary Outcome: Depression
Description: as for outcome 1
Time Frame: Post-operative (day 3)
Measure: Mean (Standard Deviation); unit: mean overall score
Arm/Group | Reiki/Manual Therapy | Usual Care Quiet Time
Number analyzed (Participants) | 136 | 136
mean overall score | 0.29 (0.41) | 0.40 (0.50)

3. Primary Outcome: Anxiety
Description: The Brief Symptom Inventory has a anxiety dimension that includes 6 items. Participants are asked to consider the "past week" when responding and each item is scored on a 5-point scale, from 0 (not at all) to 4 (extremely). The higher the score, the worse the anxiety; score range is 0-24.
Time Frame: Pre-operative (baseline)
Measure: Mean (Standard Deviation); unit: mean overall score
Arm/Group | Reiki/Manual Therapy | Usual Care Quiet Time
Number analyzed (Participants) | 136 | 136
mean overall score | 0.81 (0.77) | 0.94 (0.83)

4. Primary Outcome: Anxiety
Description: as for outcome 3
Time Frame: Post-operative (day 3)
Measure: Mean (Standard Deviation); unit: mean overall score
Arm/Group | Reiki/Manual Therapy | Usual Care Quiet Time
Number analyzed (Participants) | 136 | 136
mean overall score | 0.60 (0.60) | 0.78 (0.86)

5. Primary Outcome: Sleep
Description: The Richards-Campbell Sleep Questionnaire (RCSQ) Valid and Reliable survey with 5 domains (sleep depth, sleep latency, awakenings from sleep, ability to return to sleep, and sleep quality) and 1 question for each domain, therefore the tool has a total of 5 items.
  The visual analog scale uses statements on either side of a 0 to 100 mm horizontal line. For example, deep sleep ____ light sleep. Participants place a vertical line on the horizontal 100mm scale, to reflect which item on the scale best matches the response to each question. A ruler is used to record the mm marking of each item. A sleep score is created by dividing the sum of the length in mm of visual analog lines by 5.
  Higher scores indicates greater sleep disturbances.
Time Frame: Paper surveys distributed pre-operative (baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reiki/Manual Therapy | Usual Care Quiet Time
Number analyzed (Participants) | 136 | 136
score on a scale | 38.5 (22.2) | 39.2 (22.4)

6. Primary Outcome: Sleep
Description: as for outcome 5
Time Frame: Paper surveys distributed post-operative (day 3) after final reiki and manual therapies intervention or quiet time sessions were completed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reiki/Manual Therapy | Usual Care Quiet Time
Number analyzed (Participants) | 136 | 136
score on a scale | 42.7 (26.1) | 46.7 (25.2)

7. Primary Outcome: Pain Level, Mean Score
Description: Pain intensity was assessed on a numerical scale of 0-10 by nurses as part of usual care documentation which was generally completed every 4 hours (higher score = worst pain). Mean scores are presented as median with (P25, P75) by group
Time Frame: Post-operative thru day 3 after the 1st intervention/usual care was administered
Measure: Median (Inter-Quartile Range); unit: median and [Q1, Q3] of the mean score
Arm/Group | Reiki/Manual Therapy | Usual Care Quiet Time
Number analyzed (Participants) | 134 | 133
median and [Q1, Q3] of the mean score | 2.5 [1.7 to 3.4] | 2.5 [1.8 to 3.3]

8. Primary Outcome: Pain Level, Median Score
Description: Pain intensity was assessed on a numerical scale of 0-10 by nurses as part of usual care documentation which was generally completed every 4 hours (higher score = worst pain). Data represent median (P25, P75) score values by group.
Time Frame: Post-operative thru day 3 after the 1st intervention/usual care was administered
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Reiki/Manual Therapy | Usual Care Quiet Time
Number analyzed (Participants) | 134 | 133
score on a scale | 1.0 [0.00 to 3.0] | 1.5 [0.00 to 3.0]

9. Primary Outcome: Hospital Length of Stay, Days - Mean (Standard Deviation)
Description: Length of stay equals date of surgery (day 0) to date before the day of hospital discharge (we do NOT include the day of discharge). The number is continuous and is based on the actual length of the POSTOPERATIVE hospital stay and is based on being in the hospital at 12 MN. There is no pre-specified maximum number.
Time Frame: Days of hospital stay
Measure: Mean (Standard Deviation); unit: mean overall days and standard deviation
Arm/Group | Reiki/Manual Therapy | Usual Care Quiet Time
Number analyzed (Participants) | 136 | 136
mean overall days and standard deviation | 6.3 (2.6) | 6.5 (2.9)

10. Primary Outcome: New-onset Postoperative Atrial Fibrillation Complication
Description: Dichotomous variable (Yes versus No) based on medical record documentation of new-onset postoperative atrial fibrillation anytime in the postoperative period. The total number of "yes" responses were compared between groups as a "count".
Time Frame: Post-operation (from day of surgery until hospital discharge)
Measure: Count of Participants; unit: Participants
Arm/Group | Reiki/Manual Therapy | Usual Care Quiet Time
Number analyzed (Participants) | 136 | 136
Participants | 46 | 51

11. Primary Outcome: All-cause 30-day Hospital Readmission
Description: All-cause 30-day hospital readmission rate based on medical record data.
Time Frame: 30 days after discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Reiki/Manual Therapy | Usual Care Quiet Time
Number analyzed (Participants) | 136 | 136
Participants | 4 | 11

12. Primary Outcome: Total Opioid IV Narcotic Burden (Mean) in mg
Description: Data retrieved via a hospital billing database
Time Frame: Total opioid IV narcotic medication dose (in milligrams), using morphine equivalent data, during the length of stay, an average 6.4 days
Measure: Median (Inter-Quartile Range); unit: morphine milligram equivalents
Arm/Group | Reiki/Manual Therapy | Usual Care Quiet Time
Number analyzed (Participants) | 136 | 136
morphine milligram equivalents | 20 [10 to 31.5] | 18.4 [10 to 29.2]

13. Primary Outcome: Total Oral Narcotic Burden (Mean) in Milligarms
Description: Data retrieved via a hospital billing database
Time Frame: Total oral narcotic medication dose in milligrams, using morphine equivalent data, during the length of stay, an average 6.4 days
Measure: Median (Inter-Quartile Range); unit: morphine milligram equivalents
Arm/Group | Reiki/Manual Therapy | Usual Care Quiet Time
Number analyzed (Participants) | 136 | 136
morphine milligram equivalents | 60 [30 to 94.5] | 55.3 [30 to 87.5]

14. Secondary Outcome: Number of Participants With Hospital Re-admission Within 30 Days
Description: Number of participants with hospital re-admission within 30 days of discharge. Data retrieved medical record chart review.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Reiki/Manual Therapy | Usual Care Quiet Time
Number analyzed (Participants) | 136 | 136
Participants | 4 | 11

ADVERSE EVENTS:
Time Frame: Not applicable; the intervention, REIKI, was a NON-treatment that was not directly related to patient events that could have occurred; therefore no event data were collected.
Description: For the 0 participants at risk (e.g., All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events, were not monitored/assessed.
Arm/Group | Reiki/Manual Therapy | Usual Care Quiet Time
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-24): https://cdn.clinicaltrials.gov/large-docs/50/NCT05853250/Prot_SAP_000.pdf